CLINICAL TRIAL: NCT00025155
Title: A Phase II Evaluation of Epothilone-B BMS 247550 (NSC # 710428) in the Treatment of Recurrent or Persistent Platinum and Paclitaxel Refractory Ovarian or Primary Peritoneal Cancer
Brief Title: Ixabepilone in Treating Patients With Ovarian Epithelial or Primary Peritoneal Cancer That Has Not Responded to Previous Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02413; NCI-2012-02413 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068927; GOG-0126M (Other: Gynecologic Oncology Group); GOG-0126M (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — ixabepilone

ARMS (1):
- Treatment (ixabepilone) (Experimental): Patients receive ixabepilone IV over 1 hour. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 2 additional courses after achieving CR.
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra

SUMMARY:
Phase II trial to study the effectiveness of ixabepilone in treating patients who have recurrent or persistent ovarian epithelial or primary peritoneal cancer that has not responded to previous chemotherapy. Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of ixabepilone in patients with recurrent or persistent platinum and paclitaxel-refractory ovarian epithelial or primary peritoneal cancer.

II. Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE:

Patients receive ixabepilone IV over 1 hour. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 2 additional courses after achieving CR.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial cancer or primary peritoneal cancer

  * Recurrent or persistent disease
  * Platinum AND taxane-resistant or refractory disease

    * Progressed during therapy
    * Refractory disease within 6 months of therapy
* Measurable disease

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * Tumor lesions located within a previously irradiated field are not considered measurable disease unless there is documented tumor progression in these lesions or biopsy confirmation ≥ 90 days following completion of radiotherapy
* Ineligible for higher priority GOG (Gynecologic Oncology Group) protocol
* No active brain metastases
* Performance status - GOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT (serum glutamate oxaloacetate transaminase) ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No sensory or motor neuropathy > grade 1
* No dementia or altered mental status
* No other serious uncontrolled medical disorder
* No active infection requiring antibiotics
* No prior hypersensitivity reaction to paclitaxel or other therapy containing Cremophor EL
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 3 weeks since prior biologic therapy
* At least 3 weeks since prior immunotherapy
* Must have received:

  * 1 prior combination taxane-based and platinum-based chemotherapy regimen
  * 1 prior platinum-based chemotherapy regimen AND 1 prior taxane-based chemotherapy regimen
* Initial treatment may include high-dose therapy, consolidation, or extended therapy
* At least 3 weeks since prior chemotherapy and recovered
* No prior ixabepilone
* No other prior cytotoxic chemotherapy for recurrent or persistent disease, including treatment with initial regimen
* At least 1 week since prior hormonal anticancer therapy
* Concurrent hormone replacement therapy allowed
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to site(s) of measurable disease
* No radiotherapy to > 25% of marrow-containing areas
* Recovered from recent surgery
* At least 3 weeks since other anticancer therapy
* No prior anticancer therapy that precludes study participation
* No concurrent food supplements (e.g., St. John's wort)
* No concurrent amifostine or other protective agents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ixabepilone): Patients receive ixabepilone IV over 1 hour on days of 1, 8 and 15 of a 28-day cycle. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 2 additional courses after achieving CR.
Period: Overall Study
Arm/Group | Treatment (Ixabepilone)
Started | 51
Completed | 49 (Patients who were eligible and received any study treatment.)
Not Completed | 2
Not completed — Ineligible: Wrong primary cancer site | 1
Not completed — Ineligible: Second primary cancer site | 1

BASELINE CHARACTERISTICS:
Population: Patients who were eligible and received any study treatment.
Arm/Group | Treatment (Ixabepilone)
Number analyzed (Participants) | 49
Age, Customized [Number; unit: participants]
  20-29 years | 1
  30-39 years | 0
  40-49 years | 6
  50-59 years | 13
  60-69 years | 15
  70-79 years | 13
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 49
International Federation of Gynecology and Obstetrics (FIGO) Stage - Recurrent/Persistent [Number; unit: participants] — International Federation of Gynecology and Obstetrics, stage grouping for primary carcinoma of the ovary (1985)
  participants | 49
Histologic Type [Number; unit: participants]
  Adenocarcinoma, unspecified | 1
  Clear Cell Carcinoma | 4
  Endometrioid Adenocarcinoma | 2
  Mixed Epithelial Carcinoma | 3
  Mucinous Adenocarcinoma | 1
  Serous Adenocarcinoma | 38

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Percentage of participants with complete and partial tumor response as assessed by the Gynecologic Oncology Group Response Evaluation Criteria in Solid Tumors (GOG RECIST) with one-sided 90% Confidence Interval.
  Complete Response (CR), disappearance of all target and non-target lesions without evidence of new lesion; Partial Response (PR), >=30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD with no unequivocal progression of non-target lesions and no evidence of new lesion, or a 50% decrease in the LD in the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam with no unequivocal progression of non-target lesions and no evidence of new lesion. Complete or partial response requires confirmation at greater than or equal to 4 weeks from initial documentation.
Time Frame: Every other cycle until the completion of study treatment with an average of study treatment time as of 3 months.
Population: Eligible and treated participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ixabepilone)
Number analyzed (Participants) | 49
percentage of participants | 14.3 [8 to 100]

2. Primary Outcome: Number of People With Adverse Effects
Time Frame: Every cycle until completion of study treatment up to 30 days after stopping study treatment
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1: Number of patients who experienced a grade 1 event using Common Toxicity Criteria version 2.0
- Grade 2: Number of patients who experienced a grade 2 event using Common Toxicity Criteria version 2.0
- Grade 3: Number of patients who experienced a grade 3 event using Common Toxicity Criteria version 2.0
- Grade 4: Number of patients who experienced a grade 4 event using Common Toxicity Criteria version 2.0
Arm/Group | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4
Number analyzed (Participants) | 49 | 49 | 49 | 49 | 49
Participants
  Leukopenia | 13 | 9 | 20 | 6 | 1
  Thrombocytopenia | 39 | 10 | 0 | 0 | 0
  Neutropenia | 17 | 10 | 12 | 9 | 1
  Anemia | 9 | 23 | 13 | 4 | 0
  Hematologic | 43 | 0 | 3 | 3 | 0
  Allergy | 46 | 1 | 2 | 0 | 0
  Cardiovascular | 45 | 3 | 0 | 1 | 0
  Coagulation | 47 | 0 | 0 | 2 | 0
  Fatigue | 11 | 16 | 15 | 6 | 1
  Dermatologic | 23 | 13 | 13 | 0 | 0
  Endocrine | 48 | 1 | 0 | 0 | 0
  Gastrointestinal | 10 | 15 | 14 | 9 | 1
  Genitourinary/Renal | 41 | 6 | 1 | 1 | 0
  Hemorrhage | 48 | 1 | 0 | 0 | 0
  Hepatic | 36 | 10 | 2 | 1 | 0
  Infection | 43 | 2 | 2 | 2 | 0
  Metabolic | 36 | 6 | 3 | 4 | 0
  Neurologic | 20 | 12 | 14 | 3 | 0
  Ocular | 48 | 0 | 1 | 0 | 0
  Pain | 29 | 10 | 8 | 1 | 1
  Pulmonary | 37 | 1 | 9 | 2 | 0

3. Secondary Outcome: Progression Free Survival
Description: Progression-Free Survival is the period from study entry until disease progression, death or date of last contact, whichever occurs first.
  Progression is defined as at least a 20% increase in the sum of the longest dimensions (LD) of target lesions taking as reference the smallest sum LD recorded since study entry, or a 50% increase in the LD taking as reference the smallest LD recorded since study entry in the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, or unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions, or global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or death due to disease without prior objective documentation of progression.
Time Frame: From study entry to disease progression, death or date of last contact, whichever occurs first. Every other cycle, up to 5 years of follow-up
Population: Eligible and treated participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ixabepilone)
Number analyzed (Participants) | 49
Months | 4.4 [2.2 to 5.7]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years of follow-up.
Population: Eligible and treated participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ixabepilone)
Number analyzed (Participants) | 49
Months | 14.8 [9.9 to 17.5]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Arm/Group | Treatment (Ixabepilone)
Serious Adverse Events (participants affected / at risk) | 16/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ixabepilone) (N=49)
Anemia (Blood and lymphatic system disorders) | 1
Thrombosis Embolism (Cardiac disorders) | 2
Rigors Chills (General disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Ascites Non-Malignant (Gastrointestinal disorders) | 1
Diarrhea Without Colostomy (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
GI Other (Gastrointestinal disorders) | 1
Hypoalbuminemia (Hepatobiliary disorders) | 1
Infection Without Neutropenia (Infections and infestations) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Voice Changes/Stridor/Larynx (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ixabepilone) (N=49)
Allergic Rhinitis (Immune system disorders) | 1
Allergic Reaction (Immune system disorders) | 3
Inner Ear/Hearing (Ear and labyrinth disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 36
Transfusion Prbc's (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 42
Hypotension (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Edema (Cardiac disorders) | 4
Thrombosis Embolism (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 4
Prothrombin Time (Vascular disorders) | 2
Partial Thromboplastin Time (Vascular disorders) | 2
Fever(No Neutropenia) (General disorders) | 3
Weight Loss (General disorders) | 5
Rigors Chills (General disorders) | 1
Weight Gain(No Vod) (General disorders) | 1
Constitutional Symptoms Other (General disorders) | 1
Fatigue (General disorders) | 39
Alopecia (Skin and subcutaneous tissue disorders) | 20
Rash Desquamation (Skin and subcutaneous tissue disorders) | 6
Skin Other (Skin and subcutaneous tissue disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 6
Flushing (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Hot Flashes/Flushes (Endocrine disorders) | 2
Sense Of Smell (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 13
Flatulence (Gastrointestinal disorders) | 3
Mouth Dryness (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dyspepsia/Heartburn (Gastrointestinal disorders) | 5
Taste Disturbance (Gastrointestinal disorders) | 7
Dysphagia Esophagitis Odynophagia (Gastrointestinal disorders) | 1
Diarrhea Without Colostomy (Gastrointestinal disorders) | 21
Constipation (Gastrointestinal disorders) | 16
Mucositis Rt (Gastrointestinal disorders) | 1
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 6
Vomitting (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 22
Gi Other (Gastrointestinal disorders) | 4
Rectal Bleeding/Hematochezia (Vascular disorders) | 1
Hematuria No Vaginal Bleeding (Vascular disorders) | 2
Ggt(Gamma-Glutamyltranspeptidase) (Hepatobiliary disorders) | 2
Hepatic Other (Hepatobiliary disorders) | 1
Hypoalbuminemia (Hepatobiliary disorders) | 4
Sgot(Alt) (Hepatobiliary disorders) | 4
Sgot(Ast) (Hepatobiliary disorders) | 8
Alkaline Phosphatase (Hepatobiliary disorders) | 7
Bilirubin (Hepatobiliary disorders) | 1
Infection Without Neutropenia (Infections and infestations) | 10
Febrile With Neutropenia (Infections and infestations) | 1
Lymphatics Other (Blood and lymphatic system disorders) | 1
Lymphatics (Blood and lymphatic system disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Metabolic Other (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesmia (Metabolism and nutrition disorders) | 11
Extrapyramidal (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 3
Mood Alteration Anxiety/Agitation (Nervous system disorders) | 5
Memory Loss (Nervous system disorders) | 1
Insomnia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Mood Alteration Depression (Nervous system disorders) | 5
Neuropathy Cranial (Nervous system disorders) | 1
Neuropathy Sensor (Nervous system disorders) | 29
Neuropathy Motor (Nervous system disorders) | 2
Vision Blurred (Eye disorders) | 1
Abdominal Pain (General disorders) | 14
Pain Other (General disorders) | 5
Pain Tumor (General disorders) | 2
Neuropathic Pain (General disorders) | 1
Headache (General disorders) | 6
Pelvic Pain (General disorders) | 2
Chest Pain (General disorders) | 2
Bone Pain (General disorders) | 1
Arthralgia (General disorders) | 7
Myalgia (General disorders) | 7
Pain Rectal/Perirectal (General disorders) | 1
Voice Changes/Stridor/Larynx (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Urinary Frequency/Urgency (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Creatinine (Renal and urinary disorders) | 3
Renal/Gu Other (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Syndromes Other (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less